CLINICAL TRIAL: NCT04596267
Title: The Effects of the Histamine-3 Receptor Inverse Agonist Pitolisant on Alcohol Self-Administration in Heavy Drinkers
Brief Title: Pitolisant Effects on Alcohol Self-Administration in Heavy Drinkers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study funding was exhausted prior to reaching the recruitment goal due to pandemic related delays
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-40959; 1R21AA028864-01 (NIH)
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Use Disorder; Alcohol Drinking
Keywords: pitolisant; Wakix
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — pitolisant

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled, crossover design trial that will test the effect of pitolisant on alcohol self-administration and craving following a priming dose of alcohol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blind. Medications are over-encapsulated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pitolisant (Experimental): Subjects will take an 8.9 mg dose (two 4.45 mg pills) of pitolisant once per day on day 1 through 4. On day 5, 8.9 mg will be taken in front of staff prior to an alcohol self administration trial.
  Interventions: Drug: Pitolisant
- Placebo (Placebo Comparator): Subjects will take an placebo once per day on day 1 through 4. On day 5, a placebo will be taken in front of staff prior to an alcohol self administration trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitolisant — 8.9mg Pitolisant for 5 days
  Other Names: wakix
  Arms: Pitolisant
Drug: Placebo — Inert ingredients
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, crossover design trial that will test the effect of pitolisant on alcohol self-administration and craving following a priming dose of alcohol. The specific objective of this proposal is to determine whether pitolisant has effects on alcohol consumption and craving

DETAILED DESCRIPTION:
The present proposal is intended to answer the call for accelerating drug development by exploring the potential of a novel anticonvulsant, Pitolisant as a candidate medication for the treatment of AUD. Pitolisant is an H-3 receptor inverse agonist that is FDA-approved for treating narcolepsy which has been found to have effects of on alcohol craving and consumption in preclinical studies. The aims of this study are to test the effects of Pitolisant on alcohol self-administration and craving among a sample of non-treatment seeking heavy drinkers. The effects of 5-days of pitolisant (8.9mg) or placebo will be evaluated in a human laboratory using an alcohol self-administration methodology. In this within-subjects crossover design, heavy drinkers (N=28) will be randomized to the order of exposure (Pitolisant or placebo) prior to completing two alcohol self-administration trials. Subjects will receive a priming drink of alcohol and will have access to 8 alcoholic drinks over a 2-hour period. The investigators anticipate that subjects will consume less alcohol during an alcohol self-administration trial when receiving Pitolisant compared to when they are receiving placebo. Significant Pitolisant-induced reductions in the quantity of alcohol self-administered will be considered to be an indication that this drug may have value as an AUD medication. This study may provide a rationale for phase II clinical studies testing Pitolisant with a treatment-seeking AUD population.

ELIGIBILITY:
Inclusion Criteria:

1. 21-55 years of age
2. Able to verify age with a state or federal picture identification
3. Exceeds safe weekly drinking limits during the 28 days prior to consent (average of 14 drinks for women or 21 drinks for men per week)
4. Reports at least one episode of binge drinking (>3 drinks for women, >4 drinks for men) in the 28 days prior consent.
5. Meets DSM-5 criteria for mild alcohol use disorder or greater severity.
6. Has a smartphone to complete medication exposure period study assessments.

Exclusion Criteria:

1. Seeking treatment for alcohol problems
2. Clinical Institute Withdrawal Assessment at ≥10
3. DSM-5 diagnosis of current major depression, bipolar disorder, schizophrenia, bulimia/anorexia, dementia, insomnia disorder or a substance use disorder other than alcohol, nicotine, marijuana or caffeine
4. If female, pregnant, nursing, have plans to become pregnant
5. If female, does not agree to use an accepted form of birth control
6. Has a medical contraindication to the use of pitolisant
7. Has medical or mental condition for which further alcohol exposure at the planned dose range would be contraindicated
8. Current risk of suicidality (MINI suicidality score greater than 8 (low risk) or Yes to the ideation question #4 of the C-SSRS)
9. BMI is greater than 40 or less than 18
10. Impaired renal function (GFR <80 mL/min)
11. Have a history of any clinically significant renal or hepatic disease
12. Child-Pugh Score equal to or greater than Class B (evaluated based on presence or absence of encephalopathy and ascites, INR, bilirubin, and albumin) [https://www.mdcalc.com/child-pugh-score-cirrhosis-mortality]
13. Have a clinically significant ECG as determined by the investigator or abnormal ECG heart rate (<45 or >100 bpm) or QTc interval corrected for heart rate using the Fridericia formula (QTcF) > 450 msec
14. Have a history of cardiac arrhythmias or who for other reasons are at risk for developing Torsade de Pointes including those with bradycardia, hypokalemia, and congenital QT interval prolongation
15. Has received alcohol counseling or other non-pharmacologic intervention to treat AUD in the past 90 days
16. Has taken medications that are used to treat AUD in the past 90 days
17. Has urine toxicology results positive for cocaine, opioids, amphetamines, buprenorphine, methadone, methamphetamines, oxycontin, barbiturates, or benzodiazepines.
18. Subject is taking a medication which will significantly alter drug metabolism (e.g., strong CYP2D6 inhibitors, strong CYP3A4 inducers, or H1 receptor antagonists that cross the blood barrier (e.g. diphenhydramine or meclizine).
19. Subject is known to be a poor CYP2D6 metabolizer.
20. Subject is unable to comfortably abstain from nicotine for a period of 8 hours.
21. Has Chronic Obstructive Pulmonary Disease (COPD), history of solid organ transplant, sickle cell disease, severe heart disease or other health condition for which exposure to COVID-19 represents an unreasonable risk as determined by the study staff physician using accepted COVID-19 guidance (e.g. Centers for Disease Control, etc.).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Devine, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Psychiatry Research Center, Clinical Studies Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data from this study will be submitted to the NIAAA Data archive (https://nda.nih.gov/).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A.total of 9 subjects were enrolled and 7 completed the study.
Groups:
- Pitolisant Then Placebo: This is a within subjects design study in which each subject receives both study drug and placebo. Subjects in this group received a dose of 8.9 mg (two 4.45 mg pills) of pitolisant once daily over a 7-day period and a dose of 17.8 mg (one 17.8 mg pill) of pitolisant once daily over a 5-day period before the first alcohol self-administration trial and 12 days of matched placebo before the second alcohol self-administration trial.
- Placebo Then Pitolisant: This is a within subjects design study in which each subject receives both study drug and placebo. Subjects in this group received 12 days of matched placebo before the first alcohol self-administration trial and a dose of 8.9 mg (two 4.45 mg pills) of pitolisant once daily over a 7-day period and a dose of 17.8 mg (one 17.8 mg pill) of pitolisant once daily over a 5-day period before the second alcohol self-administration trial.
Period: Medication Dispense/Exposure Period 1
Arm/Group | Pitolisant Then Placebo | Placebo Then Pitolisant
Started | 4 | 5
Completed | 3 | 4
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Period: Alcohol Self-Administration Trial 1
Arm/Group | Pitolisant Then Placebo | Placebo Then Pitolisant
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Medication Dispense/Exposure Period 2
Arm/Group | Pitolisant Then Placebo | Placebo Then Pitolisant
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Alcohol Self-Administration Trial 2
Arm/Group | Pitolisant Then Placebo | Placebo Then Pitolisant
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitolisant Then Placebo | Placebo Then Pitolisant | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 33 (7.9) | 30.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption in Alcohol Self-Administration Trials
Description: Alcohol consumption will be measured by using a graduated cylinder to determine the amount of alcohol given to the subject that was not consumed. This outcome will be measured as standard drink units (SDU). A standard drink contains approximately 0.6 fluid ounces of pure alcohol. Lower SDUs are favorable.
Time Frame: 2.6 hours
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Total SDUs
Groups:
- Pitolisant: Subjects received 12 days of Pitolisant before the alcohol self-administration trial.
- Placebo: Subjects received 12 days of placebo before the alcohol self-administration trial.
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Total SDUs | 67.214 (25.759) | 66.786 (15.369)

2. Primary Outcome: Alcohol Consumption (BAC): Observation Period, Minute 10
Description: Alcohol consumption will be measured throughout the study by their Blood Alcohol Content (BAC) measured by a breathalyzer test. Lower BACs are favorable
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Grams of alcohol/210 Liters of breath
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Grams of alcohol/210 Liters of breath | 0.034 (0.005) | 0.033 (0.010)

3. Primary Outcome: Alcohol Consumption (BAC): Observation Period, Minute 20
Description: as for outcome 2
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Grams of alcohol/210 Liters of breath
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Grams of alcohol/210 Liters of breath | 0.038 (0.009) | 0.0364 (0.011)

4. Primary Outcome: Alcohol Consumption (BAC): Observation Period, Minute 30
Description: as for outcome 2
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Grams of alcohol/210 Liters of breath
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Grams of alcohol/210 Liters of breath | 0.037 (0.003) | 0.034 (0.009)

5. Primary Outcome: Alcohol Consumption (BAC): Observation Period, Minute 40
Description: as for outcome 2
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Grams of alcohol/210 Liters of breath
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Grams of alcohol/210 Liters of breath | 0.033 (0.006) | 0.031 (0.006)

6. Primary Outcome: Alcohol Consumption (BAC): Self-administration Block 1, Minute 30
Description: as for outcome 2
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Grams of alcohol/210 Liters of breath
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Grams of alcohol/210 Liters of breath | 0.069 (0.046) | 0.063 (0.033)

7. Primary Outcome: Alcohol Consumption (BAC): Self-administration Block 1, Minute 60
Description: as for outcome 2
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Grams of alcohol/210 Liters of breath
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Grams of alcohol/210 Liters of breath | 0.072 (0.037) | 0.047 (0.021)

8. Primary Outcome: Alcohol Consumption (BAC): Self-administration Block 2, Minute 30
Description: as for outcome 2
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Grams of alcohol/210 Liters of breath
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Grams of alcohol/210 Liters of breath | 0.086 (0.040) | 0.075 (0.046)

9. Primary Outcome: Alcohol Consumption (BAC): Self-administration Block 2, Minute 60
Description: as for outcome 2
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: Grams of alcohol/210 Liters of breath
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
Grams of alcohol/210 Liters of breath | 0.079 (0.047) | 0.082 (0.056)

10. Secondary Outcome: Alcohol Craving During 12-day Drug Exposure
Description: The Visual Analog Scale (VAS) will be used to assess alcohol craving during the medication exposure period. The VAS is a 10 cm straight line with one end meaning no alcohol craving and the other end meaning intense alcohol craving. Higher VAS scores are associated with more cravings. Lower VAS scores are favorable.
Time Frame: 12 days
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 53.2 (30.1) | 47.2 (33.7)

11. Secondary Outcome: Alcohol Consumption During the 12-day Drug Exposure
Description: Alcohol consumption during the 12 days of drug exposure will be measured using the timeline followback method. Lower (Standard Drink Units) SDUs are favorable.
Time Frame: 12 days
Population: 19 subjects were consented but 10 dropped out prior to randomization in the study (ineligible after screening or lost to follow-up). A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: SDUs
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
SDUs | 67.2 (25.8) | 66.8 (15.4)

12. Secondary Outcome: Alcohol-induced Stimulation: Observation Period, Minute 10
Description: Whether pitolisant increases the stimulant effects of a priming drink of alcohol will be assessed using the Biphasic Alcohol Effects Scale (BAES). It is a self-report, unipolar adjective rating scale that is designed to measure both stimulant and sedative effects of alcohol. It consists of fourteen items, that comprise two subscales (stimulant and sedative). Items are rated on a eleven-point scale from 0 (not at all) to 10 (extremely). The stimulant subscale can range from 0 to 70 and the sedative scale can rage from 0 to 50. Higher BAES scores are associated with more stimulant and sedative effects, respectively. This section focuses solely on stimulation. Lower BAES scores are favorable.
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 31.714 (20.878) | 30.714 (12.433)

13. Secondary Outcome: Alcohol-induced Stimulation: Observation Period, Minute 20
Description: Whether pitolisant increases the stimulant effects of a priming drink of alcohol will be assessed using the Biphasic Alcohol Effects Scale (BAES). It is a self-report, unipolar adjective rating scale that is designed to measure both stimulant and sedative effects of alcohol. It consists of fourteen items, that comprise two subscales (stimulant and sedative). Items are rated on a eleven-point scale from 0 (not at all) to 10 (extremely). The stimulant subscale can range from 0 to 70 and the sedative scale can rage from 0 to 50. Higher scores are associated with more stimulant and sedative effects, respectively. This section focuses solely on stimulation. Lower BAES scores are favorable.
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 31.429 (19.957) | 30.714 (12.433)

14. Secondary Outcome: Alcohol-induced Stimulation: Observation Period, Minute 30
Description: as for outcome 13
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 29.571 (18.183) | 31.857 (13.322)

15. Secondary Outcome: Alcohol-induced Stimulation: Observation Period, Minute 40
Description: as for outcome 13
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 29.714 (17.557) | 31.000 (14.944)

16. Secondary Outcome: Alcohol-induced Stimulation: Self-Administration Block 1, Minute 30
Description: as for outcome 13
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 32.143 (19.463) | 32.000 (11.719)

17. Secondary Outcome: Alcohol-induced Stimulation: Self-Administration Block 1, Minute 60
Description: as for outcome 13
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 31.571 (18.831) | 34.429 (14.954)

18. Secondary Outcome: Alcohol-induced Stimulation: Self-Administration Block 2, Minute 30
Description: as for outcome 13
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 31.286 (17.792) | 33.714 (15.348)

19. Secondary Outcome: Alcohol-induced Stimulation: Self-Administration Block 2, Minute 60
Description: as for outcome 13
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 28.714 (16.680) | 32.714 (16.007)

20. Secondary Outcome: Alcohol-induced Sedation: Observation Period, Minute 10
Description: Whether pitolisant increases the sedative effects of a priming drink of alcohol will be assessed using the Biphasic Alcohol Effects Scale (BAES). It is a self-report, unipolar adjective rating scale that is designed to measure both stimulant and sedative effects of alcohol. It consists of fourteen items, that comprise two subscales (stimulant and sedative). Items are rated on a eleven-point scale from 0 (not at all) to 10 (extremely). The stimulant subscale can range from 0 to 70 and the sedative scale can rage from 0 to 50. Higher scores are associated with more stimulant and sedative effects, respectively. This section focuses solely on sedation. Lower BAES scores are favorable.
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 12.714 (8.920) | 18.857 (15.742)

21. Secondary Outcome: Alcohol-induced Sedation: Observation Period, Minute 20
Description: as for outcome 20
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 9.429 (5.827) | 18.286 (14.407)

22. Secondary Outcome: Alcohol-induced Sedation: Observation Period, Minute 30
Description: as for outcome 20
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 7.286 (5.407) | 18.286 (17.114)

23. Secondary Outcome: Alcohol-induced Sedation: Observation Period, Minute 40
Description: as for outcome 20
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 8.571 (7.300) | 18.286 (17.026)

24. Secondary Outcome: Alcohol-induced Sedation: Self-Administration Block 1, Minute 30
Description: as for outcome 20
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 9.714 (7.041) | 20.714 (18.848)

25. Secondary Outcome: Alcohol-induced Sedation: Self-administration Block 1, Minute 60
Description: as for outcome 20
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 10.286 (8.440) | 18.143 (18.614)

26. Secondary Outcome: Alcohol-induced Sedation: Self-administration Block 2, Minute 30
Description: as for outcome 20
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 11.286 (10.323) | 17.571 (18.537)

27. Secondary Outcome: Alcohol-induced Sedation: Self-administration Block 2, Minute 60
Description: as for outcome 20
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 9.571 (14.316) | 16.286 (19.914)

28. Secondary Outcome: Alcohol Urge: Self-administration Block 1, Minute 30
Description: The Alcohol Urge questionnaire (AUQ) is an 8 item measure of self-reported urges to drink in human laboratory studies that assesses the participant's urge for an alcoholic drink at the time the questionnaire is completed, Questions are in the form of a 7-point Likert scale (from strongly disagree to strongly agree) and participants select the extent to which they disagree or agree with the 8 statements relating to desire to drink, expectation of a desired outcome from drinking, and inability to avoid drinking if alcohol was available. The minimum AUQ score is 8 and the maximum score is 56. Lower AUQ scores are associated with less urge for an alcoholic drink, and therefore more favorable.
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 26.57 (10.937) | 24.00 (3.964)

29. Secondary Outcome: Alcohol Urge: Self-administration Block 1, Minute 60
Description: as for outcome 28
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 23.43 (11.674) | 27.14 (11.466)

30. Secondary Outcome: Alcohol Urge: Self-administration Block 2, Minute 30
Description: as for outcome 28
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 21.29 (13.048) | 23.29 (12.079)

31. Secondary Outcome: Alcohol Urge: Self-administration Block 2, Minute 60
Description: as for outcome 28
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 4
score on a scale | 22.00 (12.055) | 22.43 (11.731)

32. Secondary Outcome: Alcohol Craving: Observation Period, Minute 10
Description: Alcohol craving will be measured by self report with the Visual Analog Scale (VAS). The VAS is a straight line with one end meaning no alcohol craving (score of 0) and the other end meaning intense alcohol craving (score of 100). The Participant marks a point on the line that matches their amount of alcohol craving. Lower VAS score is favorable.
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 44.57 (22.970) | 34.71 (21.623)

33. Secondary Outcome: Alcohol Craving: Observation Period, Minute 20
Description: as for outcome 32
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 44.43 (31.405) | 37.14 (23.398)

34. Secondary Outcome: Alcohol Craving: Observation Period, Minute 30
Description: as for outcome 32
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 47.29 (26.266) | 39.57 (26.038)

35. Secondary Outcome: Alcohol Craving: Observation Period, Minute 40
Description: as for outcome 32
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Subjects received 12 days of pitolisant before the alcohol self-administration trial.
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 50.57 (29.051) | 34.86 (25.016)

36. Secondary Outcome: Alcohol Craving: Self-administration Block 1, Minute 30
Description: as for outcome 32
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 41.29 (24.965) | 39.86 (28.962)

37. Secondary Outcome: Alcohol Craving: Self-administration Block 1, Minute 60
Description: as for outcome 32
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 42.14 (27.492) | 40.86 (31.519)

38. Secondary Outcome: Alcohol Craving: Self-administration Block 2, Minute 30
Description: as for outcome 32
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 35.00 (33.650) | 45.57 (31.133)

39. Secondary Outcome: Alcohol Craving: Self-administration Block 2, Minute 60
Description: as for outcome 32
Time Frame: 1 minute
Population: A total of 9 subjects were randomized and 7 completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 7 | 7
score on a scale | 41.14 (35.315) | 42.43 (29.860)

ADVERSE EVENTS:
Time Frame: Up to 48 Days
Description: The primary risks of this study were risks related to taking study medication, loss of confidentiality, discomfort with study procedures, overconsumption of alcohol, and interference with efforts for recovery from alcohol use disorder. These risks were adequately minimized by study design and adherence to the study protocol.
Groups:
- Pitolisant: This is a within subjects design study in which each subject receives both study drug and placebo. Subjects received a dose of 8.9 mg (two 4.45 mg pills) of pitolisant once daily over a 7-day period and a dose of 17.8 mg (one 17.8 mg pill) of pitolisant once daily over a 5-day period before the first alcohol self-administration trial.
- Placebo: This is a within subjects design study in which each subject receives both study drug and placebo. Subjects in this group received 12 days of matched placebo before the first alcohol self-administration trial.
Arm/Group | Pitolisant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 2/7 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pitolisant (N=7) | Placebo (N=7)
Bright yellow urine (Renal and urinary disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased Thirst (General disorders) | 1 (1) | 0 (0)
Left Ankle Pain (General disorders) | 1 (1) | 0 (0) — Due to sprained ankle
Right knee contusion with abrasion (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment was impacted by COVID-19 restrictions on human subject research, leading to a smaller number of subjects analyzed than planned. This study start date was also delayed due to problems securing the medication supply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT04596267/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT04596267/ICF_000.pdf